CLINICAL TRIAL: NCT01911715
Title: A Phase I Open-label Study to Investigate the Mass Balance and Biotransformation of a Single Oral 160 mg (100 µCi) Dose of 14C-MDV3100 (ASP9785) in Healthy Male Subjects
Brief Title: A Study to Explore the Routes of Elimination of MDV3100
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 9785-CL-0001; 2011-000089-37 (EudraCT Number)
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Subjects; Pharmacokinetics of MDV3100
Keywords: Phase 1; Mass Balance; MDV3100; Xtandi; Enzalutamide; Metabolism; Excretion
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Oral MDV3100 dose (Experimental)
  Interventions: Drug: MDV3100

INTERVENTIONS:
Drug: MDV3100 — Oral
  Other Names: Xtandi; enzalutamide

SUMMARY:
A study to investigate the excretion routes of radio-labelled MDV3100.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index within 18.5 to 30.0kg/m2
* Regular defecation pattern (minimum once per 2 days).
* Subject must be non-fertile, i.e., surgically sterilized or must practice an adequate contraceptive method to prevent pregnancies as defined in the protocol.

Exclusion Criteria:

* Known or suspected hypersensitivity to MDV3100, or any components of the formulation used.
* Any of the liver function tests above the upper limit of normal. A retest to confirm the result may be performed once.
* Any clinically significant history of asthma, eczema, any other allergic condition or previous severe hypersensitivity to any drug (excluding non-active hay fever).
* Abnormal pulse and/or blood pressure measurements at the pre-study visit as follows: Pulse <40 or >90 bpm; mean systolic blood pressure >140 mmHg ; mean diastolic blood pressure >90 mmHg (blood pressure measurements taken in triplicate after subject has been resting in supine position for 5 min; pulse will be measured automatically).
* A QTc interval of > 430 ms after repeated measurements (consistently after duplicate measurements), a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS).
* Use of any prescribed or OTC (over-the-counter) drugs (including vitamins, natural and herbal remedies, e.g. St. John's wort) in the 2 weeks prior to admission to the Clinical Unit, except for occasional use of paracetamol (up to 3 g/day).
* Regular use of any inducer of metabolism (e.g., barbiturates, rifampin) in the 3 months prior to admission to the Clinical Unit.
* Positive serology test for HBsAg, anti HAV (IgM), anti-HCV or anti-HIV 1+2.
* Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton (excluding spinal column)), during work or during participation in a clinical study in the previous year.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Assessment of Pharmacokinetic profile of total radioactivity in plasma and whole blood by Maximum concentration (Cmax) | Day 1 through Day 78 (21 times)
Assessment of Pharmacokinetic profile of total radioactivity in plasma and whole blood by Time to attain Cmax (tmax) | Day 1 through Day 78 (21 times)
  Time to attain Cmax (tmax)
Assessment of Pharmacokinetic profile of total radioactivity in plasma and whole blood by Time to reach quantifiable concentrations (tlag) | Day 1 through Day 78 (21 times)
Assessment of Pharmacokinetic profile of total radioactivity in plasma and whole blood by AUC from the time of dosing to the last measurable concentration (AUC0-t) | Day 1 through Day 78 (21 times)
Assessment of Pharmacokinetic profile of total radioactivity in plasma and whole blood by AUC extrapolated to infinity (AUC0-inf) | Day 1 through Day 78 (21 times)
Assessment of Pharmacokinetic profile of total radioactivity in plasma and whole blood by Terminal Disposition Rate Constant (λz) | Day 1 through Day 78 (21 times)
Assessment of Pharmacokinetic profile of total radioactivity in plasma and whole blood by Apparent terminal elimination half life (t1/2) | Day 1 through Day 78 (21 times)
Assessment of Pharmacokinetic profile of total radioactivity in plasma and whole blood by Apparent total body clearance after extra vascular dosing (CL/F) | Day 1 through Day 78 (21 times)
Assessment of Pharmacokinetic profile of total radioactivity in plasma and whole blood by Apparent volume of distribution during the terminal phase after extra vascular dosing (Vz/F) | Day 1 through Day 78 (21 times)
Assessment of Pharmacokinetic profile of total radioactivity in plasma and whole blood by blood-to-plasma ratio (Ratio Cb/p) | Day 1 through Day 78 (21 times)
Assessment of 14C recovery in urine | Day 1 through Day 78 (17 times)
Assessment of 14C recovery in feces | Day 1 through Day 78 (16 times)
Assessment of total 14C recovery (urine and feces combined) within 24 hours | Day 1 through Day 78 (17 times for urine and 16 times for feces)
Assessment of total 14C recovery (urine and feces combined) after Time of last quantifiable concentration (tlast) | Day 1 through Day 78 (17 times for urine and 16 times for feces)
Assessment of Pharmacokinetic profile of MDV3100 and metabolites in plasma | Day 1 through Day 78 (21 times)
  PK of MDV3100, MDPC0001, and MDPC0002 in plasma based on validated LC-MS/MS methods:
  * In plasma: Cmax, tmax, tlag, AUC0-t, AUC0-inf, λz, t1/2, CL/F (parent only), and Vz/F (parent only)
  The ratios of AUCMDV3100/AUC14C , AUCMDPC0001/AUCMDV3100 and AUCMDPC0001/AUC14C (and the same for MDPC0002) will be calculated
Assessment of Pharmacokinetic profile of MDV3100 and metabolites in urine | Day 1 through Day 78 (17 times)
  PK of MDV3100, MDPC0001, and MDPC0002 in urine based on validated LC-MS/MS methods:
  * In urine: Cumulative amount excreted in urine from time zero to the last measurable concentration after dosing (Ae0-t), Renal clearance (CLR), Percent of dose excreted in urine from time zero to the last measurable concentration after dosing (Ae0-t%), Cumulative amount excreted in urine from time zero extrapolated to infinity (Ae0-inf), Percent of dose excreted in urine from time zero extrapolated to infinity (Ae0-inf%)
  The ratios of AUCMDV3100/AUC14C , AUCMDPC0001/AUCMDV3100 and AUCMDPC0001/AUC14C (and the same for MDPC0002) will be calculated
Metabolic Profile: Profiling of possible metabolites of MDV3100 in plasma, urine, and feces | Day 1 through Day 78 (14 times)
  Identification and possible quantification of metabolites in plasma, and if applicable, in urine and feces

SECONDARY OUTCOMES:
Safety as assessed by recording adverse events, laboratory assessments, vital signs and electrocardiograms (ECGs) | Day 1 through Day 78

CONTACTS AND LOCATIONS:
Overall Officials: Operation Senior Research Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- PRA International, Zuidlaren, Netherlands

REFERENCES:
- [Derived] Gibbons JA, Ouatas T, Krauwinkel W, Ohtsu Y, van der Walt JS, Beddo V, de Vries M, Mordenti J. Clinical Pharmacokinetic Studies of Enzalutamide. Clin Pharmacokinet. 2015 Oct;54(10):1043-55. doi: 10.1007/s40262-015-0271-5. PMID 25917876